CLINICAL TRIAL: NCT03021577
Title: Comparison of Orbital Versus Rotational Atherectomy Effects On Coronary Microcirculation in Percutaneous Coronary Intervention (PCI)
Brief Title: Comparison of Orbital Versus Rotational Atherectomy Effects On Coronary Microcirculation in PCI
Acronym: ORACLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Jeffrey W. Moses, Professor of Cardiology in Medicine, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAQ9267
Record Dates: First submitted 2016-12-05; First posted 2017-01-16 (Estimated); Results first posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Coronary Artery Disease (CAD)
Keywords: orbital atherectomy system; rotational atherectomy; Fractional flow reserve; coronary flow reserve; index of microcirculatory resistance (IMR)
MeSH Terms: conditions — Coronary Artery Disease | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Orbital Atherectomy System (OAS) Group (Active Comparator): Subjects randomized to OAS. In a subset of patients (n= 20) a baseline cardiac magnetic Resonance Imaging (MRI) scan will be performed prior to PCI and repeated 24 hours after PCI to quantify the total volume of myocardial necrosis secondary to PCI.
  Interventions: Device: Orbital Atherectomy System (OAS); Procedure: Magnetic Resonance Imaging (MRI)
- Rotational Atherectomy (RA) Group (Active Comparator): Subjects randomized to RA using the Rotablator Rotational Atherectomy System. In a subset of patients (n= 20) a baseline cardiac magnetic Resonance Imaging (MRI) scan will be performed prior to PCI and repeated 24 hours after PCI to quantify the total volume of myocardial necrosis secondary to PCI.
  Interventions: Device: Rotablator Rotational Atherectomy System; Procedure: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Device: Orbital Atherectomy System (OAS) — The Cardiovascular Systems, Inc. (CSI) Diamondback 360 Coronary Orbital Atherectomy System (OAS) is a catheter-based system designed for facilitating stent delivery in patients with coronary artery lesions. The OAS consists of the hand-held CSI DIAMONDBACK 360 Coronary Orbital Atherectomy Device (OAD), the CSI Saline Infusion Pump (OAS pump), the CSI ViperWire Advance Coronary Guide Wire (VIPERWIRE guide wire), and the CSI ViperSlide Lubricant.
  Arms: Orbital Atherectomy System (OAS) Group
Device: Rotablator Rotational Atherectomy System — The Rotablator Rotational Atherectomy System is comprised of a Rotablator RotaGlide, a Rotablator RotaLink Plus/RotaWire/Console
  Arms: Rotational Atherectomy (RA) Group
Procedure: Magnetic Resonance Imaging (MRI) — In a subset of patients (n= 20) a baseline cardiac MRI will be performed prior to PCI and repeated 24 hours after PCI to quantify the total volume of myocardial necrosis secondary to PCI.

SUMMARY:
The investigators hypothesize that the orbital atherectomy system (OAS), a newer generation atherectomy device, reduces the incidence of microcirculatory compromise as compared to older generation rotational atherectomy (RA) due to differences in the mechanism of athero-ablation.

DETAILED DESCRIPTION:
The presence of heavily calcified coronary lesions necessitates the use of ablative devices that aid in successful percutaneous coronary intervention (PCI). However, atherectomy devices generate microparticles that embolize to the distal coronary microcirculation and may compromise myocardial tissue perfusion.

Two mechanisms that deserve particular attention are the eccentric mounting of the OAS crown and the higher flow rates on the vasodilator flush. Firstly, as opposed to rotational atherectomy where the larger, centrally mounted burr may cause obstruction of flow during the atherectomy, the smaller eccentrically mounted crown in OAS allows continuous perfusion during both atherectomy as well as rest periods. Second, both during rest and atherectomy, the flow rates of vasodilatory flush is higher in OAS compared to RA. Combined, these differences in coronary and vasodilator flush flow could lead to improved perfusion of the distal circulation, particularly during the atherectomy runs when risk of embolization is highest.

The loss of microcirculatory function can be transient, with partial or complete restoration of microcirculatory blood flow, or permanent. As shown in studies of patients with acute coronary syndromes, the loss of microcirculatory function is a critical and independent predictor of myocardial recovery and adverse outcomes. The putative protective effects of OAS on coronary microvasculature may therefore be of major clinical significance and impact.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patient with an indication for PCI including:

   * Angina (stable or unstable),
   * Silent ischemia (a visually estimated target lesion diameter stenosis of ≥70%, a positive non-invasive stress test, or FFR ≤0.80 must be present),
   * Non-ST Segment Elevation Myocardial Infarction (NSTEMI)
3. Patients will undergo cardiac catheterization and possible or definite PCI with intent to stent using any non-investigational metallic drug-eluting stent (DES)
4. Signed written informed consent
5. Heavily calcified (severe)lesions necessitating atherectomy.

Angiographic inclusion criteria:

1. The target lesion must be located in a native coronary artery with visually estimated reference vessel diameter of ≥2.25 mm to ≤4.00 mm.
2. Lesion length between 20 mm and 50mm

Exclusion Criteria:

1. Estimated creatinine clearance <30 ml/min using Cockcroft-Gault equation, unless the patient is on dialysis;
2. ST-elevation Myocardial Infarction (STEMI) within 24 hours of initial time of presentation to the first treating hospital, whether at a transfer facility or the study hospital.
3. PCI within 24 hours preceding the study procedure.
4. Cardiogenic shock (defined as persistent hypotension (systolic blood pressure <90 mm/Hg for more than 30 minutes) or requiring pressors or hemodynamic support, including intra-aortic balloon pump (IABP), at time of procedure.
5. Mobitz II second degree or complete heart block
6. Malignant ventricular arrhythmias requiring treatment
7. Pulmonary edema defined as patient with shortness of breath, evidence of volume overload on physical exam, and crepitations on physical exam (>1/3 of lungs) or radiographic interstitial or alveolar pulmonary edema
8. Subject is intubated.
9. Known left ventricular ejection fraction (LVEF) <35%.
10. Severe valvular disease (e.g. severe mitral regurgitation or severe aortic stenosis)
11. Patient is participating in any other investigational drug or device clinical trial that has not reached its primary endpoint.
12. Women who are pregnant or breastfeeding (women of child-bearing potential must have a negative pregnancy test within one week before treatment).

General Inclusion - MRI Sub-Study

1. Patients with no prior MI/scarring in the subtended myocardial territory.
2. Patients with no contraindication for MRI studies
3. Patients who could safely receive Gadolinium (i.e. estimated glomerular filtration rate (eGFR) >30)

Angiographic Exclusion Criteria:

1. Lesion length <20mm
2. Study target lesion in a bypass graft
3. Ostial right coronary artery (RCA) study target lesion
4. Chronic total occlusion (Thrombolysis In Myocardial Infarction (TIMI) flow 0/1) study target lesion
5. Bifurcation study lesion with a planned dual stent strategy
6. In-stent restenosis study target lesion

General Inclusion - MRI Sub-Study

1. Patients with no prior myocardial infarction (MI)/scarring in the subtended myocardial territory.
2. Patients with no contraindication for Magnetic resonance imaging (MRI) studies
3. Patients who could safely receive Gadolinium (i.e. eGFR>30)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2019-03-16 (Actual); Study Completion 2019-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ziad A. Ali, MD, Study Chair — Columbia University; Jeffrey W. Moses, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Orbital Atherectomy System (OAS) Group: OAS was used in percutaneous coronary intervention (PCI) of participants.
- Rotational Atherectomy (RA) Group: RA was used in percutaneous coronary intervention (PCI) of participants.
Period: Overall Study
Arm/Group | Orbital Atherectomy System (OAS) Group | Rotational Atherectomy (RA) Group
Started | 17 | 20
Completed | 17 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Orbital Atherectomy System (OAS) Group | Rotational Atherectomy (RA) Group | Total
Number analyzed (Participants) | 17 | 20 | 37
Age, Customized [Count of Participants; unit: Participants]
  ≥ 18 years | 17 | 20 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 11 | 15 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Index of Microcirculatory Resistance (IMR)
Description: Index of Microvascular Resistance (IMR) is defined as the distal coronary pressure multiplied by the hyperaemic mean transit time. IMR = Pd x Tmn at maximal hyperemia. This is for micro vascular function.
Time Frame: Up to 1 hour
Measure: Median (Inter-Quartile Range); unit: mmHg·s
Arm/Group | Orbital Atherectomy System (OAS) Group | Rotational Atherectomy (RA) Group
Number analyzed (Participants) | 17 | 20
mmHg·s | 15 [13 to 17] | 25 [14 to 53]

2. Primary Outcome: Fractional Flow Reserve (FFR)
Description: FFR is defined as the ratio of (i.e., percent of normal) flow in the stenotic artery to the flow in the same artery in the theoretic absence of the stenosis.
Time Frame: Up to 1 hour
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Orbital Atherectomy System (OAS) Group | Rotational Atherectomy (RA) Group
Number analyzed (Participants) | 17 | 20
ratio | 0.85 [0.85 to 0.88] | 0.88 [0.87 to 0.93]

3. Primary Outcome: Coronary Flow Reserve (CFR)
Description: Coronary Flow Reserve (CFR) is the ratio between hyperemic and basal coronary flow. CFR=Hyperemic Flow /Resting Flow. This is for micro vascular function.
Time Frame: Up to 1 hour
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Orbital Atherectomy System (OAS) Group | Rotational Atherectomy (RA) Group
Number analyzed (Participants) | 17 | 20
ratio | 1.9 [1.3 to 3.1] | 2.3 [1.2 to 3.7]

4. Other Pre Specified Outcome: Troponin I Level
Description: Blood test that helps determine incidence of peri-PCI myonecrosis.
Time Frame: 1 hour
Population: Data was not collected due to PI's departure from the institution following completion of data collection for the purposes of the Primary Outcome Measures.
Arm/Group | Orbital Atherectomy System (OAS) Group | Rotational Atherectomy (RA) Group
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Creatinine Kinase (CKMB) Level
Description: Blood test that helps determine incidence of peri-PCI myonecrosis.
Time Frame: 1 hour
Population: as for outcome 4
Arm/Group | Orbital Atherectomy System (OAS) Group | Rotational Atherectomy (RA) Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 18 hours post procedure.
Arm/Group | Orbital Atherectomy System (OAS) Group | Rotational Atherectomy (RA) Group
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/20
Other Adverse Events (participants affected / at risk) | 0/17 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/77/NCT03021577/Prot_SAP_002.pdf